CLINICAL TRIAL: NCT06715020
Title: Establishment and Clinical Transformation of ADC Drug Efficacy Evaluation System for Breast Cancer Based on Molecular Imaging
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Collaborators: Yunnan Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024KT104
Record Dates: First submitted 2024-11-26; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 68Ga-TTP (Experimental): All study participants will be allocated to this arm (single-arm study).Study participants will undergo 68Ga-TTP PET scans
  Interventions: Drug: 18F-FDG

INTERVENTIONS:
Drug: 18F-FDG — All study participants will undergo one 18F-FDG PET scan.

SUMMARY:
The objective of the study is to construct a noninvasive approach 68Ga-TTP PET/CT to detect the TROP2 expression of tumor lesions in patients with breast tumors and evaluate the efficacy of ADC drug therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old, male or female, ECOG score 0 or 1 points (see the table in Annex 2 for the score table);
2. Blood routine and liver and kidney function meet the following criteria: Blood routine: WBC ≥ 4.0×109 L or neutrophil ≥1.5×109 /L, PLT ≥ 100×109/L, Hb≥ 90 g/L; PT or APTT ≤ 1.5 ULN; Liver and kidney function: T-Bil ≤ 1.5×ULT(upper limit of normal), ALT and AST≤ 2.5 ULN or ≤ 5×ULT(subjects with liver metastasis), ALP ≤ 2.5 ULN(ALP ≤ 4.5 ULN if there is bone metastasis or liver metastasis); BUN ≤ 1.5×ULT, SCr ≤ 1.5×ULT;
3. Patients with confirmed or suspected breast cancer;
4. Expected survival ≥12 weeks;
5. Good follow-up compliance;
6. Women of childbearing age (15 to 49 years old) must undergo a pregnancy test within 7 days before the start of the test and the result is negative; Fertile men and women must consent to the use of effective contraception to ensure pregnancy during the study period and within 3 months of the examination;
7. Subject patients can fully understand and voluntarily participate in this experiment, and sign informed consent.

Exclusion Criteria:

1. Severe abnormal liver and kidney function;
2. Pregnant, pregnant and lactating women;
3. Can not lie flat for half an hour;
4. Unable to obtain informed consent;
5. Suffering from claustrophobia or other mental illness;
6. People who are known to be allergic to the investigational drug or its excipients in the investigational therapy;
7. Other conditions deemed unsuitable for participation in the trial by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value（SUV） | 2 years
  The uptake of the tracer （68Ga-TTP） in solid tumor lesions or suspected tumor lesions by measuring SUV on PET/CT.